CLINICAL TRIAL: NCT04840004
Title: Efficacy and Safety of PVT-1 Treatment in Patients With Advanced and Refractory Non-Small Cell Lung Cancer
Brief Title: Efficacy and Safety of PVT-1 Treatment in Patients With Advanced Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: PlusVitech S.L. (Other)
Collaborators: ECONiX Araştırma Analiz ve Danışmanlık A.Ş. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLUSV_00
Record Dates: First submitted 2021-04-05; First posted 2021-04-09 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Non Small Cell Lung Cancer; Advanced Cancer; Refractory Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PVT-1 (Other): One arm study.
  Interventions: Drug: PVT-1

INTERVENTIONS:
Drug: PVT-1 — Since there is no specific dose range is available for testing the anti-tumor effects of PVT-1 in clinical trials settings, in the present study the dose of PVT-1 will be up-titrated 250/160/160 mg to maximum 1000/640/640 mg as described in study methodology section.

SUMMARY:
Lung cancer is one of the most common causes of cancer death worldwide. It is projected that the vast majority, approximately 80% -85% of all lung cancer diagnosis is Non-Small Cell Lung Cancer (NSCLC). Although there are significant improvements in the treatment of Lung Cancer in recent years, there is still an unmet medical need for a specific population which has advanced NSCLC and mostly is refractory to existing treatments.

In NSCLC the molecular profile is important to direct the treatment. Specifically, for cases with an EGFR+, ALK+, ROS1+ or PD1/PDL1+ molecular profile, targeted treatments are available. PVT-1 is a safe, orally administrable and well-tolerated drug directed against a specific therapeutic target of cancer cells what has demonstrated efficacy in NSCLC with a molecular profile EGFR-, ALK-, ROS1- and refractory to anti-PD1 / PDL1, in last line, which also represents the highest percentage of patients and with the highest chances of cancer progression with currently available treatments.

ELIGIBILITY:
Inclusion Criteria:

Female or male with age > 18 years' old Personally signed and dated informed consent that indicating that the participant ( or a legal representative) has been informed of all aspects of the study Histologically or cytologically confirmed non-small cell lung cancer(NSCLC) NSCLC patients who are not suitable for surgery or radical radiotherapy or chemotherapy, or who have failed to or are intolerable for standard treatment in local advanced or metastatic NSCLC Diagnosis of a metastatic or locally advanced NSCLC with molecular profile EGFR (-), ALK (-) and ROS-1 (-), refractory to existing treatments Evidence of disease radiological measurable. Defined as at least one target lesion that can be accurately measured by imaging, at least one dimension as ≥20 mm with conventional computed tomography (CT), ≥10 mm with spiral CT scan (≥15mm for lymph node) Absence of untreated or symptomatic brain metastases or that requires the use of steroids.

Life expectancy of at least three months in the opinion of investigators ECOG performance status of 0-1 Time since last treatment received: 3 weeks from last QT cycle or 6 weeks if nitrosiureas, at least 2 weeks from the last RT session before the first administration of study drug (The administration of palliative radiotherapy for bone pain is allowed by any time)

Laboratory results required at the screening visit:

Neutrophils> 1500 / mm3 Haemoglobin> 9.0g / dl Platelets> 100,000 / mm3 Total bilirubin <1.5 times above the normal ranges Transaminases: AST, ALT <2 times above the normal ranges, If there are liver metastases <5 times above normal values.

Serum creatinine <1.5 times above the normal ranges Female participants childbearing potential, must have a negative pregnancy test

Exclusion Criteria:

Pregnant female patients, Breastfeeding female patients Patients unable to meet the requirements (inclusion criteria) of the study Know hypersensitivity, history of allergic or anaphylactic reaction to the drug.

ECOG performance status ≥2 Any acute, chronic or psychiatric medical condition or laboratory abnormality that may increase the risk associated with the participation or PVT-1 administration in the study or may interfere with interpretation of the results, and in judgment of the investigator, would make the participant inappropriate for entry into this study.

Current history of alcoholism or drug addiction to DSM-IV criteria within 12 months prior to screening.

Patients with major organ dysfunctions and heart disease Patients with active tuberculosis Participation in any other clinical studies (phases I - IV) within 1 month or 5 half-lives, or participation in any clinical study of drugs that could present interaction within 1 year of screening visit.

Subjects who are directly involved in the conduct of the study, and their family members, site staff members supervised by study investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-03-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Effect | 12 months
  The primary objective of this trial is to demonstrate the effect of high dose and long-term use of PVT-1 on tumor response.

SECONDARY OUTCOMES:
Progression Free Survival and Overall Survival | 12 months
  Progression free survival (PFS) and overall survival (OS). PFS will be defined as the time from the date of patients' registration to the date of the evidence of progressive disease, death due to any cause, or the last date the patient will be known to be progression-free or alive. OS will be calculated from the date of patients' registration to the date of death from any cause or the last date the patient will be known to be alive.
High Dose | 12 months
  The evaluation of plasma concentration of high doses of PVT-1 treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Sahin Lacin, Principal Investigator — Yeditepe University
Locations (4):
- Turkey (Türkiye) (4):
  - Baskent University, Adana
  - Gazi University, Ankara
  - Yeditepe University Hospital, Istanbul
  - 19 May|s University, Samsun

IPD SHARING:
Plan to Share IPD: No